CLINICAL TRIAL: NCT03325777
Title: Approach Bias Retraining to Augment Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-04-0006
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Results first posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Nicotine Dependence
Keywords: Cigarettes; Tobacco Use
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Approach Bias Retraining Group (Experimental): Individuals in this condition will receive seven sessions of ABR training in which they are instructed to approach (pull the joystick) images tilted to the right and avoid (push the joystick) images tilted to the left. They will be told that the training may weaken automatic cigarette-approach and strengthen automatic cigarette-avoidance. Furthermore, they will be told that the opposite effect will be true for the stimuli not related to cigarettes (i.e., the positive stimuli).
  Interventions: Behavioral: Approach Bias Retraining
- Control Group (Sham Comparator): Individuals in this condition will receive seven sessions of SHAM training in which they are instructed to approach (pull the joystick) images tilted to the right and avoid (push the joystick) images tilted to the left. They will be told that the purpose of the training is to improve control over these automatic tendencies and that following the training sessions, they will easily be able to push or pull the stimuli regardless of content.
  Interventions: Behavioral: SHAM Training

INTERVENTIONS:
Behavioral: Approach Bias Retraining — The Approach Avoidance Task (AAT) used for this experiment is an implicit, computerized paradigm in which participants respond to visually presented pictures on a computer screen displaying either 1) smoking-related images or 2) positive images, by pulling a joystick either towards their body (approach movement) or pushing it away from their body (avoidance movement). By pulling the joystick towards their body, the picture grows in size; by pushing the joystick away, the picture shrinks and then disappears from the screen. Participants are instructed to pull upon seeing an image tilted to the right and to push upon seeing a left-tilt image, while ignoring the image content and responding as quickly and as accurately as possible.
  Arms: Approach Bias Retraining Group
Behavioral: SHAM Training — SHAM Training
  Arms: Control Group

SUMMARY:
Tobacco use is the most preventable cause of disease, disability, and death in the United States. Standard smoking cessation care (cognitive behavioral therapy and nicotine replacement therapy), is effective in approximately 20% of the cases, clearly indicating there is substantial room for improvement.

Current work suggests that despite standard interventions, continued substance abuse may result from addictive behaviors governed partly through automatic processes that exert their influence outside conscious control. This is important from a treatment perspective, as we should develop treatments to target implicit processes.

Among a number of promising targets for intervention, cognitive biases are important to address as they have been implicated as maintenance factors for addiction. Approach bias, defined as the automatically activated action tendency to approach smoking-related stimuli, is a relatively novel cognitive bias and has been related to failed smoking cessation. A recently developed task for approach bias assessment is the Approach Bias Retraining (ABR), a computerized joystick task increasingly used to measure automatic approach tendencies in addiction research.

This clinical trial will evaluate a smoking cessation intervention that integrates standard care with approach bias retraining. Results will provide novel information regarding the potential benefits of engaging implicit cognitive biases as a means to augment traditional smoking cessation therapy. This study has the potential to help individuals attempting to quit smoking and, ultimately, provide unique information about the importance of targeting implicit processes to complement standard care.

DETAILED DESCRIPTION:
The integrated intervention involves seven weekly 60-minute therapy sessions. The each therapy session involves 15 minutes of computerized approach bias retraining and 45 minutes of individual cognitive behavioral therapy. In order to maximize adherence, the scheduling of session visits will be individualized to each participant's schedule.

During the first therapy session, the study therapist will collect relevant smoking assessments and begin orienting the participant to the joystick procedures. The therapist will explain that the joystick task is thought to affect your automatic tendencies to approach or avoid cigarettes. At this time the participant will complete the first session of approach bias retraining.

Participants will begin therapy sessions 2-6 by completing the computerized approach bias retraining task. At session 2, the therapist will then congratulate participants for deciding to quit smoking, review the positive health consequences of quitting, and express their willingness to help the participant succeed. Participants' past quit attempts will be reviewed to identify what strategies contributed to success and what factors hindered their previous attempts and a target quit date will be set for week 6. Lastly, participants will initiate self-monitoring or track each cigarette they smoke through Quit date and note situational cues for smoking (e.g. times of the day, activities while smoking).

During therapy sessions 2-5, the therapists will then assist participants in anticipating situations in their lives that will likely place them at risk for relapse, prepare them for the possibility of lapsing, and provide strategies for coping with the potential negative emotional reactions to lapsing. In addition, therapists will advise all participants to avoid or reduce drinking and advise all participants to tell their friends and family about their quit date and will discuss ways to increase social support during the quit attempt. Lastly, therapists will instruct participants in the proper use of the nicotine patch (e.g., placement of patch, use one a day, importance of not smoking while using the patch) and help them prepare for the quit day (e.g., removing all tobacco products from their environment).

At session 6, participants will initiate a quit attempt. Therapists will provide individual support for participants during this early period of abstinence. This contact will provide the opportunity for more tailored and elaborate discussions of quitting experiences and coping strategies for anticipated high-risk situations. Therapists will also reinforce success and provide support and encouragement for participants who slip and smoke and ask participants to anticipate potential challenges to remaining abstinent from smoking and discuss strategies for coping with those situations. In addition, during this session, therapists will ask participants to discuss social supports for nonsmoking, help to develop strategies for maximizing social support systems and develop participants' skills in requesting behavioral changes from others. Beginning week 6, participants will be instructed to apply one patch daily. Participants will use the full strength 21-mg patch for 6 weeks and then be instructed to taper to the 14-mg patch for the next 1 week, and then to the 7-mg patch for the remaining 1 week.

Session 7 will be the last day that the ABR task is administered. This session will focus primarily on relapse prevention. Therapists will continue with relapse prevention tactics, including provision of social support, avoiding high-risk situations, using social support from friends/co-workers, and maintaining non-smoking lifestyle changes.

Participants will be asked to come in for a brief follow-up visit at week 9, 1- month (week 10), 2-month (week 14), and 3-month (week 18). The primary function of these visits is to gather information about the participants smoking habits post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ages 18-65 capable of providing informed consent
* Willing and able to provide informed consent, attend all study visits, and comply with the protocol
* Daily smoker for at least 1 year
* Currently smoke an average of at least 5 cigarettes per day
* Report a motivation to quit smoking of at least 5 on a 10-point scale

Exclusion Criteria:

* A lifetime history of bipolar disorder, schizophrenia, psychosis, or delusional disorders; an eating disorder in the past 6 months; organic brain syndrome, mental retardation or other cognitive dysfunction that could interfere with capacity to engage in therapy; a history of substance or alcohol abuse or dependence (other than nicotine) in the last 6 months or otherwise unable to commit to refraining from alcohol use during the acute period of study participation.
* Visual or hand-motoric impairments
* Current use of nicotine replacement therapy
* Current use of any other pharmacotherapy or psychotherapy for smoking cessation not provided by the researchers during the quit attempt
* Current use of tobacco products other than cigarettes
* Insufficient command of the English language as the treatment manual is written only in English and study staff are not fluent in other languages

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via three main channels: 1) fliers and pamphlets in community-based organizations and bulletin boards; 2) social media outlets; and 3) UT Austin resources such as UT Events and digital screen ads.
Pre-assignment Details: Of all enrolled participants, 96 met inclusion criteria and were randomized into a condition group.
Period: Overall Study
Arm/Group | Approach Bias Retraining Group | Control Group
Started | 46 | 50
Completed | 37 | 38
Not Completed | 9 | 12
Not completed — Lost to Follow-up | 9 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Approach Bias Retraining Group | Control Group | Total
Number analyzed (Participants) | 46 | 50 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 50 | 96
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (10.8) | 43.3 (10.7) | 43.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 28 | 53
  Male | 21 | 22 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 40 | 45 | 85
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 41 | 42 | 83
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 46 | 50 | 96
Baseline Approach Bias [Mean (Standard Deviation); unit: units on a scale] — The approach-avoidance task (AAT) is an implicit task that measures people's behavioral tendencies to approach or avoid stimuli in the environment.
  The AAT assessment was used to calculate approach bias tendency at the start of each training session. A positive value indicates a relatively stronger avoidance tendency in response to stimuli.
  The difference in response latencies is standardized by dividing an individual's difference in reaction time by a personalized standard deviation of the latencies.
  units on a scale | 6.4 (239.2) | 139.5 (214.4) | 75.7 (235.1)

OUTCOME MEASURES:

1. Primary Outcome: Smoking Status at 3-month Follow Up
Description: The primary outcomes were 7-day point-prevalence abstinence (PPA) and prolonged abstinence (PA) at 3-month follow-up (week 18).
  PPA was defined as self-report of no smoking (not even a puff) during the previous 7 days. Failure to maintain PA at any assessment was defined as smoking on 7 consecutive days or smoking at least once each week over the last 2 consecutive weeks. PPA and PA were assessed by study staff at each appointment using sequential timeline follow-back interviews and biochemically verified by expired carbon monoxide (CO; ≤4 ppm) at each assessment as well as by saliva cotinine (≤10 ng/mL) at weeks 14 and 18.
  The outcomes in the table below show what percentage of participants remained abstinent at the 3-month follow-up.
Time Frame: 18 weeks
Measure: Number; unit: proportion abstinent
Arm/Group | Approach Bias Retraining Group | Control Group
Number analyzed (Participants) | 46 | 50
proportion abstinent | .57 | .39
Statistical Analysis 1: Comparison: Approach Bias Retraining Group vs Control Group; Test type: Superiority; p = .014, Mixed Models Analysis — a priori threshold is p<.05; Generalized Linear Mixed Models; Slope = .71, 95% CI 2-sided [.14 to 1.27], Standard Error of Mean .29

2. Secondary Outcome: Approach Bias After 7-week Intervention Phase
Description: The approach-avoidance task (AAT) is an implicit task that measures people's behavioral tendencies to approach or avoid stimuli in the environment.
  The AAT assessment was used to calculate approach bias tendency at the start of each training session. A positive value indicates a relatively stronger avoidance tendency in response to stimuli.
  The difference in response latencies is standardized by dividing an individual's difference in reaction time by a personalized standard deviation of the latencies.
Time Frame: 18 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Approach Bias Retraining Group | Control Group
Number analyzed (Participants) | 46 | 50
units on a scale | 210 (26.04) | 39 (24.86)
Statistical Analysis 1: Comparison: Approach Bias Retraining Group vs Control Group; Test type: Superiority; p < .001, Mixed Models Analysis — a priori threshold for significance was p<.05; Mean Difference (Final Values) = 172, 95% CI 2-sided [106 to 238], Standard Error of Mean 33.2

ADVERSE EVENTS:
Time Frame: 18 weeks
Arm/Group | Approach Bias Retraining Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/50
Other Adverse Events (participants affected / at risk) | 0/46 | 3/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Approach Bias Retraining Group (N=46) | Control Group (N=50)
Seizure (Nervous system disorders) | 0 | 1 — Participant had a seizure in her sleep. She was admitted to the ER in the evening and was released the next morning. She was referred to a neurologist and has no persisting health problems since the seizure.
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 | 1 — Participant reported skin irritation to Step-3 (7 mg) nicotine patches for 2-3 weeks. Participant said he moved patch around to different places as per patch protocol. Irritation would stay up to 4 days after patch was removed.
High Blood Pressure (Vascular disorders) | 0 | 1 — Participant went to ER and reported feeling dizzy. Participant was measured to have high BP at ER. Participant's doctor changed the participant's medication. Participant fully recovered.
Dizziness, Nausea, Physical Discomfort (General disorders) | 0 | 1 — Participant wore nicotine patch at 14mg for 3 days; caused dizziness, nausea, physical discomfort. Participant discontinued patch use after 3 days. Definite relationship to study intervention. Participant fully recovered.

LIMITATIONS AND CAVEATS:
This was a pilot randomized trial and thus underpowered to detect smaller effects. Second, follow-up assessment was limited to 3-months post quit attempt, and thus cannot make inferences with respect to long-term efficacy. Third, most participants were White (86.5%). An important next step in intervention development is a larger follow-up randomized clinical trial that can test the generalizability and durability of treatment effects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT03325777/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT03325777/ICF_001.pdf